CLINICAL TRIAL: NCT01153932
Title: A Phase II, Double Blind, Exploratory, Parallel-group, Placebocontrolled Clinical Study to Assess Two Dosing Regimens of GSK2402968 for Efficacy, Safety, Tolerability and Pharmacokinetics in Ambulant Subjects With Duchenne Muscular Dystrophy
Brief Title: Phase II Doubleblind Exploratory Study of GSK2402968 in Ambulant Subjects With Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114117
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2013-08

CONDITIONS: Muscular Dystrophies
Keywords: 968; muscular dystrophy; duchenne; DMD
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous regimen; 6mg/kg once weekly (Experimental): Once Weekly
  Interventions: Drug: GSK2402968; Drug: matched placebo
- Intermittent regimen; 6mg/kg twice weekly (Experimental): Twice weekly on 1st, 3rd and 5th weeks, once weekly on 2nd, 4th and 6th weeks, and no active drug on 7th to 10th week of each 10 week cycle
  Interventions: Drug: GSK2402968; Drug: matched placebo

INTERVENTIONS:
Drug: GSK2402968 — Subcutaneous injection
  Other Names: 968
Drug: matched placebo — Subcutaneous injection
  Other Names: Placebo

SUMMARY:
The purpose of this study is to determine whether GSK2402968 given as a continuous dose and as an intermittent dose is effective and safe in the treatment of Duchenne muscular dystrophy.

DETAILED DESCRIPTION:
This is a phase II, double-blind, exploratory, parallel-group, placebo-controlled clinical study in ambulant subjects with DMD resulting from a mutation that can be corrected by exon skipping induced by GSK2402968. The study aims to randomise 54 subjects. There will be 2 parallel cohorts. Each cohort will include subjects on GSK2402968 and matched placebo in a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Ambulant subjects with Duchenne muscular dystrophy resulting from a mutation in the DMD gene, confirmed by a state-of-the-art DNA diagnostic technique covering all DMD gene exons, including but not limited to MLPA (Multiplex Ligation-dependent Probe Amplification), CGH (Comparative Genomic Hybridisation) or H-RMCA (High-Resolution Melting Curve Analysis), and correctable by GSK2402968-induced DMD exon 51 skipping,
* Males, at least 5 years of age and with a life expectancy of at least 1 year
* Able to rise from floor in ≤7 seconds (without aids/orthoses),
* Able to complete the 6MWD test with a distance of at least 75m
* Receiving glucocorticoids for a minimum of 6 months immediately prior to screening, with no significant change in total daily dosage or dosing regimen for a minimum of 3 months immediately prior to screening and a reasonable expectation that total daily dosage and dosing regimen will not change significantly for the duration of the study
* QTc <450msec
* On adequate contraception
* Able to comply with and complete all protocol requirements

Exclusion Criteria:

* any additional missing exon for DMD
* Current of history of liver or renal disease or impairment
* Acute illness within 4 weeks of the first dose
* Use of prohibited meds within 6 months of fist dose
* Current participation in any other investigational clinical trial
* Positive hepatitis B surface antigen, hepatitis C antibody test, or human immunodeficiency virus (HIV) test at screening
* Symptomatic cardiomyopathy
* Children in Care

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of 2 different dosing regimens of subcutaneous GSK2402968 administered over 24 weeks in ambulant subjects with DMD | 48 weeks

SECONDARY OUTCOMES:
To assess the safety and tolerability of 2 different dosing regimens of subcutaneous GSK2402968 administered over 48 weeks in ambulant subjects | one year
To assess the PK of 2 different dosing regimens of subcutaneous GSK2402968 administered over 48 weeks in ambulant subjects with DMD | 48 weeks
To assess long term efficacy of 2 different dosing regimens of subcutaneous GSK2402968 administered over 48 weeks in ambulant subjects with DMD | one year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Australia (2):
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Parkville, Victoria
- GSK Investigational Site, Ghent, Belgium
- GSK Investigational Site, Paris, France
- Germany (2):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Essen, North Rhine-Westphalia
- GSK Investigational Site, Jerusalem, Israel
- GSK Investigational Site, Nijmegen, Netherlands
- Spain (2):
  - GSK Investigational Site, Esplugues (Barcelona)
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Voit T, Topaloglu H, Straub V, Muntoni F, Deconinck N, Campion G, De Kimpe SJ, Eagle M, Guglieri M, Hood S, Liefaard L, Lourbakos A, Morgan A, Nakielny J, Quarcoo N, Ricotti V, Rolfe K, Servais L, Wardell C, Wilson R, Wright P, Kraus JE. Safety and efficacy of drisapersen for the treatment of Duchenne muscular dystrophy (DEMAND II): an exploratory, randomised, placebo-controlled phase 2 study. Lancet Neurol. 2014 Oct;13(10):987-96. doi: 10.1016/S1474-4422(14)70195-4. Epub 2014 Sep 7. PMID 25209738